CLINICAL TRIAL: NCT03604172
Title: Neural Response to Food Stimuli: fMRI Changes Following Cognitive Behavioral Therapy for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829018; 5K23NR017209-03 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-07-27 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Binge Eating Disorder; Overweight and Obesity
Keywords: binge eating disorder; obesity; cognitive behavioral therapy
MeSH Terms: conditions — Binge-Eating Disorder; Overweight; Obesity | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): 16-week cognitive behavioral therapy intervention for binge eating disorder
  Interventions: Behavioral: Cognitive behavioral therapy
- Waitlist control (Other): 16-weeks on waitlist then participants will be provided with 16-weeks of cognitive behavioral therapy
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The cognitive behavioral therapy intervention will consist of weekly, 50-minute individual meetings for 16 weeks with a clinician trained in cognitive behavioral therapy for binge eating disorder.
  Arms: Cognitive behavioral therapy
Behavioral: Waitlist — The waitlist group will have a 16-week waitlist period. After the waitlist period, they will be offered cognitive behavioral therapy.
  Arms: Waitlist control

SUMMARY:
The purpose of this research is to conduct a randomized controlled trial (RCT) assessing the impact of CBT on neural responses to binge eating stimuli.

DETAILED DESCRIPTION:
Females with a BMI>/=25 kg/m2 and BED will be randomized to either a 16-week, one-on-one CBT intervention (n=20) or a waitlist control (WL; n=20). Both groups will have blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI) scans at baseline and after the 16-week intervention. During the scans, participants will complete the following tasks: 1) food-specific stop signal task (SST), and 2) script-driven imagery of binge foods.

ELIGIBILITY:
Inclusion Criteria:

1. Women who meet the DSM-5 criteria for BED as diagnosed by the Eating Disorder Examination Interview
2. Ages 18 to 45 years of age
3. BMI >/=25 kg/m2
4. Premenopausal
5. Able to provide informed consent
6. Right-handed
7. Eligible female patients will be:

   * Non-pregnant, evidenced by a negative urine dipstick pregnancy test
   * Non-lactating
   * Surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study
8. Understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent

Exclusion Criteria:

1. Weight > 158.8 kg (350 lbs, due to scanner weight restrictions)
2. Supine abdominal width (with arms folded above) > 70 cm or sagittal diameter > 50 cm (due to scanner dimension restrictions)
3. Pregnant or nursing (or plans to become pregnant in the next 5 months)
4. Evidence of psychiatric disorder that significantly interferes with daily living
5. Active suicidal ideation
6. Type 1 diabetes or type 2 diabetes or A1C > 6.5%
7. Use of weight loss medications or other agents known to affect body weight (e.g., oral glucocorticoids, second-generation antipsychotic medications) in the past 3 months
8. Psychiatric hospitalization within the past 6 months
9. Self-reported alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
10. Self-reported use of illicit drugs within the past 30 days
11. Presence or history of orthopedic circumstances, metallic inserts, pacemaker, claustrophobia, or other conditions that may interfere with magnetic resonance imaging
12. Loss of ≥ 10 lb of body weight within the past 3 months
13. History of (or plans for) bariatric surgery
14. Visual, auditory, or other impairment that would affect task performance
15. Epilepsy or other brain injury
16. Participation in individual psychotherapy for BED in the prior 3 months
17. Inability to attend treatment and lack of capacity to provide informed consent
18. Any serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariana M Chao, PhD, CRNP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chao AM, Agarwal K, Zhou Y, Grilo CM, Gur RC, Joseph P, Shinohara RT, Richmond TS, Wadden TA. Neural Responses to Auditory Food Stimuli Following Cognitive Behavioral Therapy for Binge-Eating Disorder. Int J Eat Disord. 2024 Sep;57(9):1911-1923. doi: 10.1002/eat.24244. Epub 2024 Jul 2. PMID 38953334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8) | 30 (8) | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 14 | 12 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Binge eating [Mean (Standard Deviation); unit: episodes in past 4 weeks] | 13 (1) | 13 (1) | 13 (1)
Reward-based eating [Mean (Standard Deviation); unit: units on a scale] | 38 (2) | 35 (2) | 37 (8)
Disinhibition [Mean (Standard Deviation); unit: units on a scale] | 14 (1) | 13 (1) | 13 (2)

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level-dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Response to Food-specific Stop-signal Task
Description: BOLD fMRI (neural) response to high-calorie food cues during the food-specific stop-signal task in reward regions of interest. Reward-regions included BOLD response of the combination of prefrontal cortex, orbitofrontal cortex, insula, ventral tegmental area, and ventral striatum
Time Frame: Change from baseline to 16 weeks
Population: Fewer participants had usable data for the fMRI analysis than the overall trial.
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Number analyzed (Participants) | 18 | 16
percent signal change | -0.4 (0.1) | -0.3 (0.1)

2. Primary Outcome: Blood Oxygen Level-dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Response to Binge-eating Script-driven Imagery
Description: BOLD fMRI response to descriptions of binge eating episodes during script-driven imagery (contrast in reward-regions of interest between food vs neutral stimuli). Reward-regions included combination of BOLD response in the prefrontal cortex, orbitofrontal cortex, insula, ventral tegmental area, and ventral striatum.
Time Frame: Change from baseline to 16 weeks
Population: Fewer participants had usable data for the fMRI analysis than the overall trial.
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Number analyzed (Participants) | 18 | 16
percent signal change | -0.2 (0.1) | -0.3 (0.2)

3. Secondary Outcome: Binge Eating Episodes
Description: Change in number of episodes measured from the Eating Disorder Examination Questionnaire. Higher values indicate more episodes.
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: episodes in the past 28 days
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Number analyzed (Participants) | 20 | 20
episodes in the past 28 days | -9 (2) | -4 (2)

4. Secondary Outcome: Reward-based Eating Drive
Description: Change measured from the Reward-Based Eating Drive Scale. Range of 0-52 with higher scores indicting higher reward-based eating drive.
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale | -15 (3) | 3 (3)

5. Secondary Outcome: Dietary Disinhibition
Description: Self-report measured from the Eating Inventory Questionnaire. Score range of 0-16. Higher scores indicate higher levels of disinhibited eating.
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale | -4 (1) | 0 (1)

ADVERSE EVENTS:
Time Frame: Baseline to end of intervention (16 weeks)
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03604172/Prot_SAP_000.pdf